CLINICAL TRIAL: NCT00912860
Title: A Multicenter, Open-Label Immunogenicity and Safety Study of a Serum-Free Pre-Formulated Solution of AVONEX (Interferon Beta-1a) Administered Intramuscularly to Patients With Relapsing/Remitting Multiple Sclerosis
Brief Title: Immunogenicity and Safety Study of Serum-Free Avonex
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Biogen Idec MD, Biogen Idec
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: C-867
Record Dates: First submitted 2009-06-02; First posted 2009-06-03 (Estimated); Last update posted 2009-06-10 (Estimated); Status verified 2009-06

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; interferon beta-1a; avonex
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interferon beta-1a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): serum-free avonex given IM
  Interventions: Drug: Interferon beta-1a

INTERVENTIONS:
Drug: Interferon beta-1a — serum free Avonex given IM once a week
  Other Names: Avonex

SUMMARY:
To evaluate the immunogenicity of a serum-free pre-formulated solution of Avonex when given to interferon beta naive patients with relapsing/remitting multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Must have a diagnosis of relapsing/remitting MS as defined by McDonald, et al15; criteria numbers 1-4.
* Must have an expanded disability status scale (EDSS) score between 0 and 5.5, inclusive.
* Must be able to understand and comply with the protocol.

Exclusion Criteria:

* Has experienced a relapse within 2 months prior to Day 1. Relapses are defined as new or recurrent neurologic symptoms not associated with fever or infection, lasting at least 48 hours, and accompanied by new objective neurological findings upon examination by the investigator.
* History of any significant cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, and/or other major disease that would preclude therapy with interferon beta.
* Abnormal screening or baseline blood tests determined to be clinically significant by the investigator
* History of a seizure within 3 months prior to Day 1.
* History of suicidal ideation within 3 months prior to Day 1 or an episode of severe depression within 3 months prior to Day 1.
* Known allergy to natural rubber latex.

Other inclusion and exclusion criteria apply as per protocol

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 155 (Actual)
Dates: Start 2003-01; Primary Completion 2004-12 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the immunogenicity of a serum-free pre-formulated solution of AVONEX® | Study duration is 20 months

SECONDARY OUTCOMES:
To evaluate the safety of a serum-free pre-formulated solution of AVONEX® | The study duration is 20 months

CONTACTS AND LOCATIONS:
Overall Officials: Biogen-Idec Investigator, Principal Investigator — Biogen